CLINICAL TRIAL: NCT01401127
Title: A Comparison of Metabolism During Moderate Exercise Between Healthy Volunteers and People With T1DM Treated With CSII Using 70% of Their Usual Insulin Basal Rate
Brief Title: Managing Insulin Pumps for Exercise - Study 1
Status: Completed | Type: Observational
Sponsor: Buckinghamshire Healthcare NHS Trust (Other)
Collaborators: Animas Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: RXQ404(1)
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Exercise; Continuous Subcutaneous Insulin Infusion; CSII; Insulin Pump Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All samples retained will be plasma samples. Any samples remaining after analysis will be retained until the 3 trials in this research study have been completed, and will then be destroyed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 Diabetes: Participants with type 1 Diabetes running their insulin pump at 70% of usual basal rate
- Participants without diabetes: Participants without diabetes or evidence of impaired glucose regulation

SUMMARY:
People with Type 1 Diabetes Mellitus (T1DM) like to take part in sport and exercise, but problems with metabolism and blood glucose control can make this difficult. Some people with T1DM administer their insulin via an insulin pump, also know as continuous subcutaneous insulin infusion (CSII) therapy, in which a background or basal level of insulin is constantly infused under the skin by a special pump, with bolus doses of insulin given to accompany food. Clinical experience suggests that this may be particularly useful for managing diabetes for exercise, but there is limited experimental evidence to support this. The aim of this research , which is divided into three parts, is to investigate the hypothesis that the physiological response to sub-maximal (moderate) exercise of a person with type 1 diabetes treated with CSII, can be made to approximate more closely to the physiological response of a healthy individual by a prior reduction of their basal insulin infusion rate. This first part of the research is designed to compare metabolic response to exercise between people without diabetes and people with T1DM running there insulin pump at the usual basal rate.

DETAILED DESCRIPTION:
For the first part of the study, participants will be either people with type 1 diabetes treated with insulin pump therapy or volunteers without diabetes. The 2 groups will be matched as far as possible by age, body mass index and usual level of activity. Participants will attend an exercise laboratory on 2 occasions. On the first occasion, which can take place at any time of day, formal written consent will be obtained for participation in the study. Participants will then undergo measurement of maximal exercise capacity (VO2 MAX). On the second occasion they will attend 2 hours after a lunch containing 60 grams of carbohydrate (advice will be given on how this can be achieved). A cannula will be inserted on arrival and blood samples obtained. Arterialised samples will be obtained by using a heated hand technique. Once the cannula has been inserted participants with type 1 diabetes will be asked to reduce the basal insulin infusion rate on their insulin pump to 70% of normal until the end of the study visit. After 30 minutes a further set of blood samples will be obtained, and participants will then start to exercise for 1 hour at 50% VO2 MAX. A further set of blood samples will be obtained at the end of the hour of exercise. Participants will then rest for 30 minutes before a final set of blood samples is taken. At this point the cannula will be removed and the study visit ends. Participants with diabetes will be given the choice to return basal insulin infusion rate to normal at this point. A snack will be offered.

Blood glucose will be monitored every 10 minutes and also if a participant feels symptoms of hypoglycaemia. If hypoglycaemia occurs the protocol will be stopped and carbohydrate given until the blood glucose level returns to the normal range.

ELIGIBILITY:
Inclusion Criteria:

For participants with Type 1 Diabetes Mellitus

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged between 18 and 65 years
* Diagnosed with Type 1 diabetes mellitus
* Treated with CSII for at least 3 months
* Exercises regularly for more than 1 hour per week

For participants without Type 1 Diabetes Mellitus

* Participant is willing and able to give informed consent for participation in the study
* Male or female, aged between 18 and 65 years
* Exercises regularly for more than 1 hour per week

Exclusion Criteria:

For participants with type 1 Diabetes Mellitus

* People with any one of the following complications of diabetes:

  1. stage 2+ diabetic retinopathy
  2. renal impairment (with creatinine >150micromol/l)
  3. known history or symptoms of cardiovascular disease
  4. foot ulceration
  5. peripheral vascular disease
* Known pregnancy or breastfeeding
* Untreated or unstable respiratory disease
* Known hypoglycaemia unawareness
* Treatment with drugs known to interfere with glucose metabolism

For participants without Type 1 Diabetes Mellitus

* Known pregnancy or breastfeeding
* Untreated or unstable respiratory disease
* Diagnosis of impaired fasting glucose, impaired glucose tolerance or diabetes mellitus
* Treatment with drugs known to interfere with glucose metabolism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with Type 1 Diabetes treated with insulin pump therapy who exercise for at least 1 hour each week and comparable participants without diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Glucose excursion | Glucose will be measured at the start and end of 1 hour of exercise at 50% VO2 MAX during the second study visit
  The primary outcome measure is change in blood glucose (glucose excursion) between the start and the end of exercise

SECONDARY OUTCOMES:
Comparison between the two groups of levels of lactate | Samples will be obtained on arrival, 30 minutes later (at the start of exercise), at the end of exercise (1 hour later) and at the end of the study visit (30 minutes later)
Multiple correlation between blood glucose values and values of lactate, NEFA, betahydroxybutyrate, catecholamines, glucagon, insulin, C-peptide, human growth hormone and cortisol | Samples will be obtained on arrival, 30 minutes later (at the start of exercise), at the end of exercise (1 hour later) and at the end of the study visit (30 minutes later)
Ratio of respiratory quotient (RQ) at the beginning of exercise to RQ at the end of exercise, compared between the two groups, which will give information about fuel use during exercise. | Respiratory quotient will be calculated using a breath by breath analyser using 2 minutes of data from the start at the end of exercise
Comparison between the two groups of levels of non-esterified fatty acids (NEFA) | Samples will be obtained on arrival, 30 minutes later (at the start of exercise), at the end of exercise (1 hour later) and at the end of the study visit (30 minutes later)
Comparison between the two groups of levels of beta-hydroxybutyrate | Samples will be obtained on arrival, 30 minutes later (at the start of exercise), at the end of exercise (1 hour later) and at the end of the study visit (30 minutes later)
Comparison between the two groups of levels of circulating catecholamines | Samples will be obtained on arrival, 30 minutes later (at the start of exercise), at the end of exercise (1 hour later) and at the end of the study visit (30 minutes later)
Comparison between the two groups of levels of glucagon | Samples will be obtained on arrival, 30 minutes later (at the start of exercise), at the end of exercise (1 hour later) and at the end of the study visit (30 minutes later)
Comparison between the two groups of levels of circulating insulin | Samples will be obtained on arrival, 30 minutes later (at the start of exercise), at the end of exercise (1 hour later) and at the end of the study visit (30 minutes later)
Comparison between the two groups of levels of human growth hormone | Samples will be obtained on arrival, 30 minutes later (at the start of exercise), at the end of exercise (1 hour later) and at the end of the study visit (30 minutes later)
Comparison between the two groups of levels of cortisol | Samples will be obtained on arrival, 30 minutes later (at the start of exercise), at the end of exercise (1 hour later) and at the end of the study visit (30 minutes later)

CONTACTS AND LOCATIONS:
Overall Officials: Ian W Gallen, MD FRCP, Principal Investigator — Buckinghamshire Healthcare NHS Trust
Locations (1):
- Wycombe Hospital, High Wycombe, Buckinghamshire, United Kingdom